CLINICAL TRIAL: NCT04309292
Title: Dietary Protein and Skeletal Muscle in Older Twins - Targeting the Gut Microbiome to Overcome Anabolic Resistance: The PROMOTe Study
Brief Title: Protein and Skeletal Muscle in Older Twins: Role of the Gut Microbiome
Acronym: PROMOTe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1234
Record Dates: First submitted 2020-02-05; First posted 2020-03-16 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2021-02

CONDITIONS: Sarcopenia; Frailty; Age-Related Sarcopenia
Keywords: gut microbiome; metabolome; prebiotic
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): protein supplementation plus prebiotic supplementation
  Interventions: Dietary Supplement: Prebiotic food supplement; Dietary Supplement: Protein supplement
- Placebo Arm (Placebo Comparator): Protein supplementation plus placebo
  Interventions: Dietary Supplement: Protein supplement; Dietary Supplement: Maltrodextrin (placebo)

INTERVENTIONS:
Dietary Supplement: Prebiotic food supplement — Darmocare Pre = trade name Gut microbiome modulator
  Arms: Treatment Arm
Dietary Supplement: Protein supplement — commercially available protein supplementation with high leucine content
Dietary Supplement: Maltrodextrin (placebo) — Starchy substance
  Arms: Placebo Arm

SUMMARY:
Research Question: Does the gut microbiome contribute to muscle anabolic resistance to protein supplementation in older adults?

Background: Loss of muscle occurs with age and skeletal muscle in older adults can display anabolic resistance to protein in diet. It has been hypothesised that the gut microbiome may play a role in this relationship and therefore could be targeted.

Aim:

This trial aims to test whether modulation of the gut microbiome, in addition to protein supplementation, can improve skeletal muscle function versus protein supplementation alone.

Methods:

Double blinded, randomised, placebo controlled, dietary intervention study. Twin pairs will be randomised to either receive protein supplementation plus placebo or protein supplementation plus a gut microbiome modulator (prebiotic plus probiotic) for 12 weeks. Primary outcome will be muscle function measured using chair-rise time.

Conclusion:

Anabolic resistance warrants further characterisation to guide future therapeutic interventions, especially considering its role in the development of disability, sarcopenia and frailty.

DETAILED DESCRIPTION:
Research Question: Does the gut microbiome contribute to muscle anabolic resistance to protein supplementation in older adults?

Background: Loss of skeletal muscle mass and strength occurs with increasing age and is associated with loss of function, disability, and the development of sarcopenia and frailty. Dietary protein is essential for skeletal muscle function, but older adults do not respond as well as younger people to protein, so called 'anabolic resistance'. The aetiology and molecular mechanisms for this are not understood, however a number have been proposed. The gut microbiome is known to play a key role in a number of these postulated mechanisms. This has led us to hypothesise that the gut microbiome may mediate anabolic resistance and could represent an exciting new target for ameliorating muscle loss in older adults.

Aim:

This trial aims to test whether modulation of the gut microbiome, in addition to protein supplementation, can improve skeletal muscle function versus protein supplementation alone.

Methods:

Double blinded, randomised, placebo controlled, dietary intervention study. Volunteers will be recruited in twin pairs from TwinsUK cohort, for which extensive baseline data are available. The twin nature of the study allows for close genetic and environmental matching at baseline. Each pair will be randomised to either receive protein supplementation plus placebo or protein supplementation plus a gut microbiome modulator (prebiotic plus probiotic). Intervention period will be 12 weeks. Clinical and biochemical measures will be taken at 0, and 12 weeks, with 2-monthly contact. Gut microbiota composition will be measured, alongside a battery of physical assessments. Primary outcome will be muscle function measured using chair-rise time. The trial will be delivered remotely using video calls, and postal boxes.

Conclusion:

Anabolic resistance warrants further characterisation to guide future therapeutic interventions, especially considering its role in the development of disability, sarcopenia and frailty. Therapeutic options are badly needed, particularly for older adults who cannot undertake exercise programmes.

ELIGIBILITY:
Inclusion Criteria:

* Aged >=60 years
* Dietary protein intake of <1.3g/kg/day
* Able to consent
* Able to access video calls on a device such as laptop/tablet

Exclusion Criteria:

* Severe food allergy
* Current or recent antibiotic use (preceding 3 months)
* Currently or recent use of protein or leucine supplements (preceding 3 months)
* Currently or recent use of probiotic or prebiotic food supplements (preceding 3 months)
* Current or prior history of gastrointestinal disease e.g. gastrointestinal cancer, inflammatory bowel disease, bariatric surgery, irritable bowel syndrome
* history of any significant injury or surgery which currently affects physical functioning and ability to undertake chair stand test
* weight loss of ≥5% of body weight in preceding 6-12 months
* Currently involved in other intervention studies
* Any condition or circumstance likely to interfere with the normal conduct of the study and interpretation of the results, as judged by the investigators As the study population are over 60 years old, it is assumed that there will be no pregnant women who are eligible to take part.

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Change in chair rise time | baseline and end of study (12 weeks)
  Chair rise time refers to the time it takes to complete 5 chair rises, without using arms. It is a well-recognised proxy marker of muscle strength. The change from baseline chair rise time at 12 weeks is the primary outcome. The residuals of change will be used in analysis.

SECONDARY OUTCOMES:
Gripstrength, as measured by dynamometer | baseline and end of study (12 weeks)
  A marker of muscle strength, measured in kilograms. Dominant hand will be used. (absolute and change from baseline at 12 weeks)
Microbiome composition | baseline and end of study (12 weeks)
  faecal samples analysed for their microbial composition, aka the presence of bacteria in the stool. The bacteria present will be identified where possible and quantified. The diversity of the microbiota present will be calculated using standard protocols. (absolute and change from baseline at 12 weeks)
Metabolites in serum | baseline and end of study (12 weeks)
  Serum samples analysed for their metabolite composition, aka the presence of metabolites in the blood. Those present will be identified where possible and quantified. (absolute and change from baseline at 12 weeks)
Cognition | baseline and end of study (12 weeks)
  CANTAB Battery. (absolute and change from baseline at 12 weeks)
Questionnaire measures: appetite as measured by SNAQ | baseline and end of study (12 weeks)
  SNAQ: Simplified Nutritional Appetite Questionnaire (absolute and change from baseline at 12 weeks)
Questionnaire measures: physical activity as measured by IPAQ | baseline and end of study (12 weeks)
  IPAQ: international physical activity questionnaire. (absolute and change from baseline at 12 weeks)
Salivary microbiome | baseline and end of study (12 weeks)
  saliva samples analysed for their microbial composition, aka the presence of bacteria in the saliva. The bacteria present will be identified where possible and quantified. The diversity of the microbiota present will be calculated using standard protocols. (absolute and change from baseline at 12 weeks)
Urinary microbiome | baseline and end of study (12 weeks)
  Urine samples analysed for their microbial composition, aka the presence of bacteria in the urine. The bacteria present will be identified where possible and quantified. The diversity of the microbiota present will be calculated using standard protocols. (absolute and change from baseline at 12 weeks)
Anthropological measures: height | baseline and end of study (12 weeks)
  height, measured in centimetres. (absolute and change from baseline at 12 weeks)
Anthropological measures: weight | baseline and end of study (12 weeks)
  measured in kilograms. (absolute and change from baseline at 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Steves, Principal Investigator — The Department of Twin Research & Genetic Epidemiology
Locations (1):
- Department of Twin Research and Genetics, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Please see attached document DTR_DataAccess_Policy_0318.pdf for our Data Access Policy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after the study has been completed and all results analysed. We estimate this to be approximately 2023. The data will remain available for the foreseeable future with no end date in sight at present.
Access Criteria: Please see attached document DTR_DataAccess_Policy_0318.pdf for our Data Access Policy.
URL: https://twinsuk.ac.uk/wp-content/uploads/2018/11/DTR_DataAccess_Policy_0318.pdf

REFERENCES:
- [Background] Ni Lochlainn M, Bowyer RCE, Steves CJ. Dietary Protein and Muscle in Aging People: The Potential Role of the Gut Microbiome. Nutrients. 2018 Jul 20;10(7):929. doi: 10.3390/nu10070929. PMID 30036990
- [Derived] Ni Lochlainn M, Bowyer RCE, Moll JM, Garcia MP, Wadge S, Baleanu AF, Nessa A, Sheedy A, Akdag G, Hart D, Raffaele G, Seed PT, Murphy C, Harridge SDR, Welch AA, Greig C, Whelan K, Steves CJ. Effect of gut microbiome modulation on muscle function and cognition: the PROMOTe randomised controlled trial. Nat Commun. 2024 Feb 29;15(1):1859. doi: 10.1038/s41467-024-46116-y. PMID 38424099
- [Derived] Ni Lochlainn M, Nessa A, Sheedy A, Horsfall R, Garcia MP, Hart D, Akdag G, Yarand D, Wadge S, Baleanu AF, Whelan K, Steves C. The PROMOTe study: targeting the gut microbiome with prebiotics to overcome age-related anabolic resistance: protocol for a double-blinded, randomised, placebo-controlled trial. BMC Geriatr. 2021 Jul 1;21(1):407. doi: 10.1186/s12877-021-02301-y. PMID 34210274